CLINICAL TRIAL: NCT06570434
Title: A Phase 1b/2a Open Label Dose Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Budoprutug in Adult Participants With Sys-temic Lupus Erythematosus (SLE)
Brief Title: Phase 1b/2a in SLE With Budoputug
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was never initiated
Sponsor: Tenet Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ELM-119-001
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Systemic Lupus Erythematosus; SLE; B Cells
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental): Low dose
  Interventions: Drug: budoprutug
- Dose 2 (Experimental): Middle dose
  Interventions: Drug: budoprutug
- Dose 3 (Experimental): High Dose
  Interventions: Drug: budoprutug

INTERVENTIONS:
Drug: budoprutug — monoclonal antibody

SUMMARY:
The purpose of the study is to determine the safety, tolerability, and pharmacokinetics of budoprutug in participants with SLE

DETAILED DESCRIPTION:
This is a Phase 1b/2a, multicenter, open-label study designed to evaluate the safety, tolerability, PK, and PD of budoprutug in adult participants with SLE.

In Phase 1b, participants who fulfill the 2012 Systemic Lupus International Collaborating Clinics(SLICC) classification criteria for SLE, and who have active SLE (as defined by a SLEDAI ≥ 4 at Screening and Day 1),have failed at least 1 line of treatment, and who are assessed as appropriate for the study by the Eligibility Adjudicator, will be enrolled in sequential escalating dose cohorts. Three dose cohorts are planned.

The Phase 2a expansion cohort will include approximately 16 to 20 participants with active SLE, at least one-half of whom will have renal involvement. Participants will continue to be followed through Week 52 for safety, PK, and PD assessmentsParticipants will also be monitored during this time for ongoing clinical response, safety parameters, and kinetics of re-population of B-cell subsets after the return of B cells to baseline values.

ELIGIBILITY:
Inclusion Criteria:.

* Diagnosis of SLE fulfilling SLICC criteria or 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) criteria at least 24 weeks prior to study entry, with one of the following at Screening
* If taking a corticosteroid regimen prior to Screening, currently receiving ≤ 20 mg prednisone or equivalent by Day -28. Exceptions for patients with active LN are detailed in Section XX (where we talk about CS use).
* Female participants of non-childbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before the Screening Visit) or postmenopausal, defined as spontaneous amenorrhea for at least 1 year, with follicle-stimulating hormone in the postmenopausal range at Screening, as per central laboratory reference range.

Additional criteria for Phase 2a participants only:

* Hybrid SLEDAI ≥ 6 at Screening AND Day 1. Note: only the clinical aspects of hybrid SLEDAI must be confirmed on Day 1; laboratory values that contribute to hybrid SLEDAI do not need to be re-measured prior to dosing on Day 1. Additional criteria for contributions to hybrid SLEDAI are as follows:
* Participants with neurological system contribution to hybrid SLEDAI will not be enrolled.
* At least 6 points from the hybrid SLEDAI score must be derived from organ system involvement excluding points from oral ulcers, alopecia, or anti-dsDNA auto-antibododies

Additional criteria for Phase 2a participants with LN:

* Diagnosis of International Society of Nephrology/Renal Pathology Society (ISN/RPS) 2003 Class III or IV LN as evidenced by renal biopsy performed within 2 years prior to or during Screening, either with or without the presence of Class V LN.
* Proteinuria (UPCR > 1.0 gram per gram [g/g]), based on a sample from a 24 hour urine collection during Screening.
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2 (as calculated by the Chronic Kidney Disease Epidemiology Collaboration formula).
* Currently receiving 1 or more immunosuppressive agents that has been stable for dose and route of administration for ≥ 8 weeks prior to baseline.

Exclusion Criteria:

* Use of IV, intramuscular, intra-articular, or high-potency intralesional corticosteroids within 6 weeks prior to Screening or expectation of requiring parenteral corticosteroids during the study. Exceptions include protocol required pre-medication prior to infusion of budoprutug.
* Use of high-potency topical corticosteroid and/or topical agents (immunosuppressant) for skin lesions within 7 days prior to Screening
* The following laboratory values:

  * Absolute neutrophil count < 1.0 × 109/L.
  * White blood cell count < 2.0 × 109/L.
  * Cluster of differentiation (CD) 19 B-cell count <80 cells/µL.
  * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2 × ULN.
  * Total bilirubin > 1.5 × ULN, unless due to Gilbert's syndrome.
* History of serious or significant infusion reaction associated with rituximab, belimumab, anifrolumab, or other monoclonal antibody therapy.
* History of or current diagnosis of active tuberculosis, untreated latent tuberculosis infection (LTBI) or undergoing current treatment for untreated LTBI
* History of chronic (i.e., chronic urinary tract infection), recurrent (3 or more of the same type of infection in a 52-week period), latent, or recent serious infection
* Any previous use of CD19 targeted therapy (e.g., inebilizumab or cell therapy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse events (AEs) and Serious Adverse events (SAEs) | Day 1 through Week 24
  Safety assessments of budoprutug include changes in vital signs, clinical findings on physicial exam, electrocardiogram and clinical laboratory findings

SECONDARY OUTCOMES:
PK parameters | Day 1 through Week 24
  Area under the maximum observed concentration (AUC)
PK parameters | Day 1 through Week 24
  Peak concentration (Cmax)
PK parameters | Day 1 through Week 24
  Time to maximum observed concentration(T-max)
PK parameters | Day 1 through Week 24
  Terminal half-life
PK parameters | Day 1 through Week 24
  Apparent clearance
PK parameters | Day 1 through Week 24
  Volume of distribution
Immunogenicity | Day 1 through Week 24
  Incidence of anti-drug antibodies (ADA)
Immunogenicity | Day 1 through Week 24
  Time-course of anti-drug antibodies (ADA)
Immunogenicity | Day 1 through Week 24
  Titers of anti-drug antibodies (ADA)

OTHER OUTCOMES:
Exploratory | Day 1 through Week 24
  Change in urine protein creatinine ratio measured in g/g
Exploratory | Day 1 through Week 24
  Changes in b cell subsets measured in µL
Exploratory | Day 1 through Week 24
  Change over time in Physician's Global Assessment of Disease Activity
Exploratory | Day 1 through Week 24
  Change in Systemic Lupus Erythematosus Disease Activity Index
Exploratory | Day 1 through Week 24
  Change in Functional Assessment of Chronic Illness Therapy
Exploratory | Day 1 through Week 24
  Change in Participant's Global Assessment of Disease Activity

IPD SHARING:
Plan to Share IPD: No